CLINICAL TRIAL: NCT05127018
Title: Dose Higher Doses of Botulinum Toxin Show Better Intensity and Duration in the Treatment of Gummy Smile
Brief Title: Higher Doses of Botulinum Toxin in the Treatment of Gummy Smile
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Gong Xi, DDS, principal investigator, Peking University
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: pkusshighdose
Record Dates: First submitted 2021-11-09; First posted 2021-11-19 (Actual); Results first posted 2023-04-26 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Smiling; Botulinum Toxins, Type A
Keywords: gummy smile; botulinum toxin; dose
MeSH Terms: conditions — Smiling

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- the average-dose method (Active Comparator): With the average-dose method, the dose was individualized according to the severity of anterior gingival exposure pretreatment. For mild gingival smile (3-5 mm), a single-site injection of 2 U botulinum toxin type A [total, 4 U] at both the right and left levator labii superioris alaeque nasi muscles) was administered. For moderate (5-7 mm) and severe (≥7 mm) gingival smile, 3 U and 5 U of botulinum toxin type A, respectively, were injected per side (total, 6 U and 10U, respectively). The injection points were located at bilateral levator labii superioris alaeque nasi muscles and at the Yonsei point26, with half doses administered at each point.
  Interventions: Drug: injection of Botulinum type A
- the higher-dose method (Experimental): With this method, patients were administered botulinum toxin type A after 8 months when the effect of the previous injection had vanished. The injection dose (U) per side was set as the absolute value of the preoperative anterior gingival exposure (mm). For example, if the preoperative anterior gingival exposure was 5mm, then the patient would be injected with 5 U of botulinum toxin per side (total, 10U). The injection points were located at bilateral levator labii superioris alaeque nasi muscles and at the Yonsei point26, with half doses administered at each point.
  Interventions: Drug: injection of Botulinum type A

INTERVENTIONS:
Drug: injection of Botulinum type A — The participates were allocated to two different application methods: Simplified Method for the first injection and Individualized Method 8 months later. All the patients underwent twice injection with each methods with no change of the BTX-A(Botox, Allergan, Irvine, CA) and other injection details: Lyophilized 100 U of Botox was reconstituted in 2.5 mL of 0.9% sodium chloride solution. The injections were made with a 27-gauge insulin syringe. The treatment was an outpatient procedure and all injections were performed by one of the authors (X.G.). No anesthesia was given during the procedure.
  Other Names: injection of Botulinum type A(Botox, Allergan, Irvine, CA)

SUMMARY:
Botulinum type A (BTX-A) is an easy and efficacious treatment for gingival smile (GS). However, the necessary for higher-doses among patients are controversial. The objective was to compare the reduction of gingival exposure using two methods in patients with different dosage. In this prospective self-controlled study, healthy GS participates who had an anterior gingival exposure (GE) of more than 3 mm were enrolled and administered with 2-5 U BTX-A (total, 4-10 U) injections into 1-2 points according to the severity presented pretreatment in the Average-dose Method. And after 8 months, the Higher-doses Method was administered the same point injection of 3-10 U BTX-A (total, 6-20 U). Data were collected at baseline and 4, 12, 32 and 60 weeks of follow-up.

DETAILED DESCRIPTION:
The smile is one of the universal facial expressions of humans. Gingival smile is characterized by gingival exposure of >3 mm upon smiling. The degree of gingival exposure can vary substantially between patients, with patients presenting gingival exposure of up to more than 10 mm. The prevalence of gingival smile is 10.57%, and it is more frequently observed in females. Although gingival smile is merely an anatomical variation, it can be considered unattractive, causing significant distress and impacting one's quality of life. Moreover, most orthodontists and dentists regard gingival smile as an important risk factor for dental treatment.

Gingival smile involves a complex interaction between the facial muscles, bone, and skin; specifically, it is related to hypermobility of the upper lip with muscle involvement and alterations in anatomical features, such as a short clinical dental crown, anterior dentoalveolar extrusion, maxillary excess, and a short upper lip. Therapies for gingival smile range from botulinum toxin injections to surgical interventions according to its etiology. Although the outcomes of surgical procedures are long-lasting, botulinum toxin type A treatment is an easy and fast outpatient procedure that requires no downtime and has high efficacy rates. Nevertheless, there are controversies around the optimal dose and injection site of botulinum toxin type A. Moreover, the efficiency of botulinum toxin type A for gingival smile varies markedly between studies, with the improvement rate of gingival exposure ranging from 62.06% to 98%. Sucupira and Abramovitz advocate the use of a low amount of botulinum toxin type A of 1.95 U per side for the treatment of gingival smile. They noted an average satisfaction level of 9.75 on a 10-point scale with this approach. They claimed that higher doses does not provide further benefit, and, in fact, could lead to lip ptosis, asymmetry, and excessive upper lip length. However, Polo disagreed with their argument, claiming 2-5 U injection of botulinum toxin type A according to the severity of gingival smile. In this regard, Garcia and Fulton showed that low-dose injection of botulinum toxin per muscle (2-5 IU) was as effective as higher doses. Though prior studies have demonstrated a correlation between higher doses of botulinum toxin and intensity and duration of muscle paralyses, no conclusion can be drawn regarding duration and intensity of doses used in the recent studies. A safe approach advocated by some authors consists of starting with low toxin doses initially, with retouching at a later stage if required. In this study, the investigators compared botulinum toxin type A efficiency using the average-dose method (2-5 U botulinum toxin type A per side determined according to the severity of anterior gingival smile) and , the higher-dose method (3-10 U botulinum toxin type A per side determined according to the severity of anterior gingival smile). The investigators aimed to assess the efficiency and duration of these approaches, as well as side effects and patients' satisfaction with treatment.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 3.0-mm anterior gingival exposure upon unrestricted, "full-blown" smiling
* healthy adults

Exclusion Criteria:

* contraindication of BTX-A
* previous diseases or treatments affecting the position of the gingiva or upper lips
* history of BTX-A injections to the head or neck region
* facial paralysis
* having received and/or receiving active orthodontic treatment that includes vertical dimension treatment, such as extrusion and intrusion, and presence of
* periodontal disease
* subject's refusal to participate

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2019-11-20 (Actual); Primary Completion 2020-08-20 (Actual); Study Completion 2021-10-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Xi Gong, Principal Investigator — Peking University School of Stomatology
Locations (1):
- Peking University School and Hospital of Stomatology, Beijing, Beijing Municipality, China

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: According to the estimated sample size, 33 participants need to be included in the study, and 33 people were actually included, but this study was a prospective, self-controlled clinical study, which is two treatments for the same group of patients, so the total sample size is 33 people.
Groups:
- The Treatment Group: In this prospective self-controlled study, healthy participants with gummy smile underwent two treatment methods. First, participants were injected with the average-dose, which the dose was individualized according to the severity of anterior gingival exposure pretreatment. For mild gingival smile (3-5 mm), a single-site injection of 2 U botulinum toxin type A [total, 4 U] at both the right and left levator labii superioris alaeque nasi muscles) was administered. For moderate (5-7 mm) and severe (≥7 mm) gingival smile, 3 U and 5 U of botulinum toxin type A, respectively, were injected per side (total, 6 U and 10U, respectively). The injection points were located at bilateral levator labii superioris alaeque nasi muscles and at the Yonsei point, with half doses administered at each point.
  And 8 months later All the patients underwent second injection of the higher-dose method.
  With this method, patients were administered botulinum toxin type A after 8 months when the effect of the previous injection had vanished. The injection dose (U) per side was set as the absolute value of the preoperative anterior gingival exposure (mm). For example, if the preoperative anterior gingival exposure was 5mm, then the patient would be injected with 5 U of botulinum toxin per side (total, 10U). The injection points were located at bilateral levator labii superioris alaeque nasi muscles and at the Yonsei point, with half doses administered at each point.
Period: the Average-dose Period
Arm/Group | The Treatment Group
Started (With the average-dose method, the dose was individualized according to the severity of anterior gingival exposure pretreatment.) | 33
Completed | 33
Not Completed | 0
Period: the Higher-dose Method Period
Arm/Group | The Treatment Group
Started (With this method, patients were administered botulinum toxin type A after 8 months when the effect of the previous injection had vanished. The injection dose (U) per side was set as the absolute value of the preoperative anterior gingival exposure (mm).) | 33
Completed | 33
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | The Treatment Group
Number analyzed (Participants) | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 33
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.1 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 2
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  China | 33
anterior gingival exposure [Mean (Standard Deviation); unit: mm] | 6.4 (1.5)

OUTCOME MEASURES:

1. Primary Outcome: Anterior Gingival Exposure (GE) 4 Weeks Post-injection
Description: The distance from the superior margin point of the right incisor to the lower margin of the upper lip upon maximum smile.
Time Frame: 4 weeks postinjection
Measure: Mean (Standard Deviation); unit: mm
Groups:
- the First Injection(the Average-dose Method): With the average-dose method, the dose was individualized according to the severity of anterior gingival exposure pretreatment. For mild gingival smile (3-5 mm), a single-site injection of 2 U botulinum toxin type A [total, 4 U] at both the right and left levator labii superioris alaeque nasi muscles) was administered. For moderate (5-7 mm) and severe (≥7 mm) gingival smile, 3 U and 5 U of botulinum toxin type A, respectively, were injected per side (total, 6 U and 10U, respectively). The injection points were located at bilateral levator labii superioris alaeque nasi muscles and at the Yonsei point26, with half doses administered at each point.
  injection of Botulinum type A: The participates were allocated to two different application methods: Simplified Method for the first injection and Individualized Method 8 months later. All the patients underwent twice injection with each methods with no change of the BTX-A(Botox, Allergan, Irvine, CA) and other injection details: Lyophilized 100 U of Botox was reconstituted in 2.5 mL of 0.9% sodium chloride solution. The injections were made with a 27-gauge insulin syringe. The treatment was an outpatient procedure and all injections were performed by one of the authors (X.G.). No anesthesia was given during the procedure.
- the Second Injection(the Higher-dose Method): With this method, patients were administered botulinum toxin type A after 8 months when the effect of the previous injection had vanished. The injection dose (U) per side was set as the absolute value of the preoperative anterior gingival exposure (mm). For example, if the preoperative anterior gingival exposure was 5mm, then the patient would be injected with 5 U of botulinum toxin per side (total, 10U). The injection points were located at bilateral levator labii superioris alaeque nasi muscles and at the Yonsei point26, with half doses administered at each point.
  injection of Botulinum type A: The participates were allocated to two different application methods: Simplified Method for the first injection and Individualized Method 8 months later. All the patients underwent twice injection with each methods with no change of the BTX-A(Botox, Allergan, Irvine, CA) and other injection details: Lyophilized 100 U of Botox was reconstituted in 2.5 mL of 0.9% sodium chloride solution. The injections were made with a 27-gauge insulin syringe. The treatment was an outpatient procedure and all injections were performed by one of the authors (X.G.). No anesthesia was given during the procedure.
Arm/Group | the First Injection(the Average-dose Method) | the Second Injection(the Higher-dose Method)
Number analyzed (Participants) | 33 | 33
mm | 3.6 (1.5) | 3.0 (1.5)

2. Secondary Outcome: Anterior Gingival Exposure (GE) 12 Weeks Post-injection
Description: as for outcome 1
Time Frame: 12 weeks postinjection
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | the First Injection(the Average-dose Method) | the Second Injection(the Higher-dose Method)
Number analyzed (Participants) | 33 | 33
mm | 5.4 (1.6) | 4.9 (1.5)

3. Secondary Outcome: Anterior Gingival Exposure (GE) 24 Weeks Post-injection
Description: as for outcome 1
Time Frame: 24 weeks postinjection
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | the First Injection(the Average-dose Method) | the Second Injection(the Higher-dose Method)
Number analyzed (Participants) | 33 | 33
mm | 6.3 (1.4) | 5.8 (1.2)

4. Secondary Outcome: Anterior Gingival Exposure (GE) 48 Weeks Post-injection
Description: as for outcome 1
Time Frame: 48 weeks postinjection
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | the First Injection(the Average-dose Method) | the Second Injection(the Higher-dose Method)
Number analyzed (Participants) | 33 | 33
mm | 7.0 (1.4) | 6.5 (1.0)

ADVERSE EVENTS:
Time Frame: For follow-up of the first injection, the participants was followed up at 4, 12 weeks and 48 weeks. For the re-injection, the participants was followed up at 4, 12, 48 weeks.
Description: The intervention in this study is low-dose injection of botulinum toxin (6U/person), which is very safe, with no participants at risk for Serious Adverse Events or for All-Cause Mortality.
Groups:
- the First Injection（the Average-dose Method）: With the average-dose method, the dose was individualized according to the severity of anterior gingival exposure pretreatment. For mild gingival smile (3-5 mm), a single-site injection of 2 U botulinum toxin type A [total, 4 U] at both the right and left levator labii superioris alaeque nasi muscles) was administered. For moderate (5-7 mm) and severe (≥7 mm) gingival smile, 3 U and 5 U of botulinum toxin type A, respectively, were injected per side (total, 6 U and 10U, respectively). The injection points were located at bilateral levator labii superioris alaeque nasi muscles and at the Yonsei point26, with half doses administered at each point.
  injection of Botulinum type A: The participates were allocated to two different application methods: Simplified Method for the first injection and Individualized Method 8 months later. All the patients underwent twice injection with each methods with no change of the BTX-A(Botox, Allergan, Irvine, CA) and other injection details: Lyophilized 100 U of Botox was reconstituted in 2.5 mL of 0.9% sodium chloride solution. The injections were made with a 27-gauge insulin syringe. The treatment was an outpatient procedure and all injections were performed by one of the authors (X.G.). No anesthesia was given during the procedure.
- the Second Injection（the Higher-dose Method）: With this method, patients were administered botulinum toxin type A after 8 months when the effect of the previous injection had vanished. The injection dose (U) per side was set as the absolute value of the preoperative anterior gingival exposure (mm). For example, if the preoperative anterior gingival exposure was 5mm, then the patient would be injected with 5 U of botulinum toxin per side (total, 10U). The injection points were located at bilateral levator labii superioris alaeque nasi muscles and at the Yonsei point26, with half doses administered at each point.
  injection of Botulinum type A: The participates were allocated to two different application methods: Simplified Method for the first injection and Individualized Method 8 months later. All the patients underwent twice injection with each methods with no change of the BTX-A(Botox, Allergan, Irvine, CA) and other injection details: Lyophilized 100 U of Botox was reconstituted in 2.5 mL of 0.9% sodium chloride solution. The injections were made with a 27-gauge insulin syringe. The treatment was an outpatient procedure and all injections were performed by one of the authors (X.G.). No anesthesia was given during the procedure.
Arm/Group | the First Injection（the Average-dose Method） | the Second Injection（the Higher-dose Method）
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/33
Other Adverse Events (participants affected / at risk) | 5/33 | 4/33
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | the First Injection（the Average-dose Method） (N=33) | the Second Injection（the Higher-dose Method） (N=33)
Slight lip ptosis (Skin and subcutaneous tissue disorders) | 5 (5) | 4 (4) — patients felt slight lip ptosis at 1-2 weeks after injection, which disappeared within 4 weeks without further intervention.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-20): https://cdn.clinicaltrials.gov/large-docs/18/NCT05127018/Prot_SAP_000.pdf